CLINICAL TRIAL: NCT02589873
Title: A Workplace Intervention Trial Comparing Two Diabetes Prevention Programs - In-person and Online - Delivered in a Large Urban Workplace Environment.
Brief Title: Getting in Balance: A Workplace Diabetes Prevention Intervention Trial
Acronym: GIBW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CN-15-2318-H
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 2; Overweight; Obesity
Keywords: Lifestyle Intervention; Workplace; Diabetes Prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- In-Person Diabetes Prevention Program (Active Comparator): An in-person group delivery modality of a CDC recognized Diabetes Prevention Program (DPP), delivered by the Young Men's Christian Association (YMCA). This group receives lifestyle coaching in a group setting, meeting weekly for 16 weeks followed by 3 biweekly sessions, and 5 monthly maintenance sessions.
  Interventions: Behavioral: In-Person Diabetes Prevention Program
- Online Diabetes Prevention Program (Active Comparator): An online delivery modality of a CDC recognized Diabetes Prevention Program (DPP), delivered by Canary Health's Virtual Lifestyle Management program. This group completes online learning sessions weekly for 16 weeks followed by 8 monthly maintenance sessions.
  Interventions: Behavioral: Online Diabetes Prevention Program

INTERVENTIONS:
Behavioral: In-Person Diabetes Prevention Program — Lifestyle intervention program involving group-based educational sessions, diet and physical activity tracking, and weekly weigh ins. Participants complete the intervention over 12 months.
  Other Names: YMCA DPP
  Arms: In-Person Diabetes Prevention Program
Behavioral: Online Diabetes Prevention Program — Lifestyle intervention program involving web-based educational videos, diet and physical activity tracking, and recording weight. Participants complete the intervention over 12 months.
  Other Names: Virtual Lifestyle Management
  Arms: Online Diabetes Prevention Program

SUMMARY:
This study evaluates two group-based Diabetes Prevention Program (DPP) lifestyle interventions delivered in the workplace to individuals at risk for pre-diabetes: 1) an in-person group-based lifestyle intervention; and 2) an internet-based intervention delivered using an online platform with lifestyle coaching support. Eligible participants will be randomized equally to each intervention program (120 participants in each).

DETAILED DESCRIPTION:
The study seeks to compare weight loss, changes in physical activity and dietary fat intake, and participant engagement in two Diabetes Prevention Program (DPP) interventions derived from the Centers for Disease Control and Prevention (CDC) curriculum: an in-person and an internet-based intervention program.

We hypothesize that the internet-based intervention will be more effective in achieving weight loss than the in-person intervention, given its convenience for participants to complete sessions and therefore greater potential engagement in the program.

ELIGIBILITY:
Inclusion Criteria:

* Ethnicity: All ethnic groups;
* Sex: all genders;
* Age (as of date of enrollment): Lower age limit: 18 years; Upper age limit: NONE;
* Body mass index ≥ 25.0 kg/m2; ≥23 kg/m2 if Asian
* Having pre-diabetes based on a score of 9+ on the CDC pre-diabetes screener
* Able and willing to enroll and provide written, informed consent, i.e., to:
* meet the time and data collection requirements of the study;
* be randomized to one of the two intervention programs;
* adhere to the recommendations of the study intervention as assigned; and
* participate in follow-up for 12 months.

Exclusion Criteria:

* Does not work at one of the participating employer work locations/departments;
* Inability to speak, read, or understand English;
* No regular access to a computer with internet capabilities;
* Diagnosis of Type 1 or Type 2 diabetes mellitus;
* Systolic blood pressure ≥ 180 mm Hg or diastolic blood pressure ≥ 100 mm Hg on more than one occasion during the last year;
* Having a medical or physical condition that make moderate intensity physical activity (like a brisk walk) difficult or unsafe, such as exercise induced asthma or chronic obstructive pulmonary disease (COPD);
* Use of weight-loss medications in the past 3 months;
* Regular use (> 5 days/month) of medications that affect appetite or weight (e.g., oral corticosteroids, insulin, oral hypoglycemics etc.);
* Currently enrolled in a weight loss program;
* Planning to undergo bariatric surgery during the study period;
* Heart disease (angina, heart attack (myocardial infarction), congestive heart failure (CHF)), stroke;
* Renal insufficiency;
* Diagnosis of cancer (other than non-melanoma skin cancer) that was active or treated with radiation or chemotherapy within the past 2 years;
* Pregnant, lactating or planning to become pregnant during the study period;
* Already enrolled or planning to enroll in a research study that would limit full participation in this study or confound the observation and interpretation of the study's findings;
* Planning to transfer to another department location during the study period;
* Planning to move out of the area during the study period;
* Investigator discretion for clinical safety or protocol adherence reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2015-09; Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Body weight lost | 12 months
  Percentage of body weight lost and the amount of weight lost (in pounds) on average over the 12 month follow-up, and at 6 and 12 months compared to baseline, by intervention arm. Body weight will be collected at baseline, 6 months, and 12 months.

SECONDARY OUTCOMES:
Change in minutes of physical activity | 12 months
  Change in physical activity duration per week - measured using the International Physical Activity Questionnaire (IPAQ);
Change in dietary fat intake | 12 months
  Change in daily dietary fat intake - measured using the Block Fat Screener
Participant engagement | 12 months
  Participant engagement - measured by the number of intervention sessions completed by 6 months, as well as the number of maintenance sessions completed between 6 and 12 months.
Stress and well-being | 12 months
  Change in well-being - measured using SF-8 Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Assiamira Ferrara, MD, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- City and County of San Francisco, San Francisco, California, United States